CLINICAL TRIAL: NCT01673880
Title: A Single-center, Open-label, Randomized, Multi-cohort, Crossover Study of Relative Bioavailability of Tablet Versus Capsule Formulation of E2006 in Healthy Adult Subjects
Brief Title: Open-Label Study of Bioavailability of E2006 Tablet Versus Capsule Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E2006-A001-005
Record Dates: First submitted 2012-08-22; First posted 2012-08-28 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-03

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

ARMS (3):
- E2006 2.5 mg (Other)
  Interventions: Drug: E2006
- E2006 10mg (Other)
  Interventions: Drug: E2006
- E2006 25 mg (Other)
  Interventions: Drug: E2006

INTERVENTIONS:
Drug: E2006 — 2.5 mg, 10 mg, and 25 mg E2006 tablets

SUMMARY:
This is a single-center, open-label, randomized crossover study being conducted in three cohorts of healthy adult subjects. Approximately 36 subjects will be randomized to one of three cohorts (approximately 12 subjects per cohort) and they will receive both a single dose of E2006 in capsule formulation and a single dose of E2006 in tablet formulation, in random sequence, at a 1:1 ratio. The doses to be tested will be 2.5 mg, 10 mg, and 25 mg.

ELIGIBILITY:
Inclusion:

* Healthy males or females,
* ages 18 to 55 years
* Body mass index (BMI) >
* 18 and 32 kg/m2 at Screening

Exclusion:

* Female subjects who are nursing
* Subjects with a history of gastrointestinal surgery (hepatectomy, nephrectomy, digestive organ resection, etc.) that may affect PK profiles of E2006
* Subjects with a known history of clinically significant drug or food allergies
* Subjects with a known allergy or hypersensitivity to capsule or tablet ingredients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of E2006 of tablet vs. capsule formulations | up to 336 hours post-dose

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Laurent, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, LLC, Austin, Texas, United States